CLINICAL TRIAL: NCT00206570
Title: Double Blind Study of Estradiol Plus Neuroleptic Versus Placebo Plus Neuroleptic in the Treatment of Psychotic Symptoms in Women With Schizophrenia
Brief Title: Clinical Estradiol Trial in Women With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Stanley Medical Research Institute (Other); National Health and Medical Research Council, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APRC 75/02; ERE-IND-INP-GRA; 143654; 00-105
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Gender differences; Hormones; Estradiol; PANSS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Estradiol

INTERVENTIONS:
Drug: Estradiol

SUMMARY:
To investigate the 'estrogen-protection' hypothesis by comparing changes in psychotic symptoms between one group of patients receiving standard antipsychotic drug treatment plus placebo and a second matched group receiving standard antipsychotic drug treatment plus 100microgram estradiol patch in a double blind controlled trial.

Hypothesis : That the women receiving adjunctive estradiol will demonstrate a more rapid and more substantial decrease in psychotic symptoms over the course of the study than the women receiving adjunctive placebo.

DETAILED DESCRIPTION:
BACKGROUND:

Schizophrenia is a severe mental disorder that affects up to two percent of the adult population. Patients present with a variety of symptoms including hallucinations, delusions and bizarre behaviour while some develop additional "negative" symptoms such as amotivational states and poverty of thought. Schizophrenia is generally thought to be an organic brain disorder with psychosocial determinants for course and outcome. The illness appears to be heterogenous with groups of patients presenting with distinct and differing patterns of psychopathology and illness course. Part of this heterogeneity includes distinct male and female subtypes of schizophrenia.

In recent times, gender differences in schizophrenia have received some attention, in particular from an epidemiological and psychopathological perspective. Hormonal studies have been utilised to investigate underlying neuroendocrine disturbances in schizophrenia, but information from these studies has not been used in the development of new gender specific treatment strategies. Overall the treatment of schizophrenia has remained gender-blind. The main gender differences observed in schizophrenia that have international consensus include the later age of onset in women, better response to neuroleptics in women, and more treatment resistant negative symptoms in men. Women have also demonstrated vulnerability to psychotic episodes during menopause, the post-partum period and at low estrogen phases of the menstrual cycle.

From these clinical observations, Seeman and Lang hypothesised that estrogen may provide "protection" against early onset of severe schizophrenia in women, thereby accounting for increased vulnerability during both lifetime and monthly low estrogen phases. Findings from both basic and clinical research warrant further investigation of the hypothesis that estrogen has a protective effect in women not only over the female life cycle, but also over the menstrual cycle.

We have been conducting clinical trials in patients with schizophrenia using estrogen as a treatment for many years, and have an international reputation for work in this area. Initially, we conducted an open clinical trial with acutely ill schizophrenic women and added 0.02mg of oral estradiol to the antipsychotic drug treatment of 11 women. Their response was compared to seven women who received antipsychotic drugs alone. The estrogen adjunct group showed dramatic earlier improvement, with significant reduction in positive psychotic symptoms by day 3 of treatment. This suggests that estradiol may act as a catalyst for treatment and could prove to be an important adjunctive treatment in the therapy of schizophrenia. Subsequent to this early pilot study, we conducted a double blind placebo controlled 3-arm study of 100mcg, 50mcg estradiol and placebo transdermal adjunctive patches. Published in Schizophrenia Research(2001), our results showed that the 100mcg estradiol adjunct afforded the best outcomes.

RESEARCH OBJECTIVES:

To investigate the usefulness of estradiol as an adjunctive treatment in schizophrenia ,by comparing changes in psychopathology between one group of patients receiving standard antipsychotic drug treatment plus a placebo skin patch and a second matched group receiving standard antipsychotic drug treatment plus a 100mcg estradiol patch in a double blind, 28 day, controlled trial.

ETHICS REVIEW AND INFORMED CONSENT:

The protocol for this study has been approved by the Alfred Ethics Committee.

Only patients who are able to give informed consent, i.e. able to demonstrate an understanding of the objectives of the study and the implications of their role in it, will be recruited into the study. Patients who are extremely psychotic or disturbed will not be approached to enter the study. Involuntary patients who are able to give informed consent will be able to participate and where possible a guardian or relative will be contacted and notified of the patients' involvement. Patients will be advised that their participation is voluntary and that they are free to withdraw from the study at any stage.

CONFIDENTIALITY:

Patients' identity will remain anonymous at all times. Once a patient agrees to participate in the study, she will be assigned a code number to ensure anonymity. Information about the subject will be restricted to the researchers directly involved, unless there are clear management issues, in which case the information will be shared with the treatment team. Patients' files will be stored in locked filing cabinets with access available to researchers only. All test results will be shared with the patient and family / guardian.

STUDY POPULATION:

A target number of 100 patients will be recruited over a three-year period with equal numbers being allocated to each group. Patients will be recruited from both inpatient and outpatient settings and patients may be recruited from other centres providing that approval has been gained from the appropriate controlling bodies.

INCLUSION CRITERIA:

Female patients who have a current DSM 4 diagnosis of Schizophrenia, Schizoaffective or Schizophreniform Disorder.

EXCLUSION CRITERIA:

* Female patients who are pregnant or lactating.
* Female patients with postpartum psychosis or related disorder
* Female patients with known abnormalities in the hypothalamo-pituitary gonadal-axis, thyroid dysfunction, central nervous system tumours.
* Female patients taking estrogen preparations such as the oral contraceptive pill.
* Female patients whose psychotic illness is directly due to illicit drugs or who have a history of substance abuse or dependence during the last 6 months.

Females with any significant unstable medical illness such as cardiovascular disease, renal disease, Addisons disease, thromboembolic disorders, epilepsy, diabetes etc.

- Post-menopausal or pre-menarche female patients.

WITHDRAWAL CRITERIA:

Patients are free to withdraw from the study at any stage without offering an explanation.

Patients experiencing any adverse effects which, in the opinion of the investigator, are serious (i.e. life threatening, requiring hospitalisation or medical treatment) will be withdrawn from the study immediately. All patients withdrawn will be followed up until the adverse event has resolved.

STUDY TREATMENTS CONCOMITANT TREATMENTS:

All patients will participate in standard in-patient and outpatient psychosocial therapies and activities as advised by their treatment team. All patients will receive psychotropic and non-psychotropic medications as per their treatment teams orders. All medications received during the study will be recorded to be included in the analysis.

STUDY MEDICATION:

The study involves the addition of transdermal 100mcg estradiol (or transdermal placebo- inactive substance) to standard antipsychotic treatment for 4 weeks. The length of the trial is 1 menstrual cycle, which is a short period of estrogen use. Most side effects commonly associated with estrogen use are related to long term administration and are thus not applicable in this study.

STUDY MEASUREMENTS:

The PANSS (Kay et al. 1987) will be performed at screening/baseline and at each evaluation visit. The PANSS consists of a Positive Scale (7 positive symptom constructs), a Negative Scale (7 negative symptom constructs) and a General Psychopathology Scale (16 symptom constructs). This scale will be the primary outcome measure of the trial.

In addition to the PANSS, the Adverse Symptom Checklist, Abnormal Involuntary Movement Scale, Simpson Angus Scale and serum hormone measurements will be completed at each visit. Cognitive testing will be performed monthly. Participants will be assessed at baseline, day 7, day 14, day 21 and day 28.

DATA MANAGEMENT:

All data gathered will be entered in the patients file under the patients code number. Files will be stored in the research unit in locked filing cabinets. Data entered on computer will be done so using the patients code number for identification. A separate booklet will be used to record data collected at screening, baseline, and evaluation visits. All files will be retained by the hospital for a period of 15 years after completion or discontinuation of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of potential child-bearing age (Pre-menopausal and Post-menarche)
* Female patients who have a current diagnosis of Schizophrenia, Schizophreniform Disorder, or Schizoaffective Disorder (not in manic phase)
* Female patients who score more than or equal to 60 on PANSS rating scale
* Female patients who are able to give informed consent

Exclusion Criteria:

* Female patients who are pregnant or lactating.
* Female patients with known severe abnormalities in the hypothalamo-pituitary gonadal axis, thyroid dysfunction, central nervous system tumours, or other serious medical conditions which would contraindicate estrogen use.
* Female patients already taking estrogen preparations such as the oral contraceptive pill
* Post-menopausal or pre-menarche female patients.
* Female patients whose psychotic illness is due to illicit drugs or who have a history of consistent substance abuse or dependence during the last 6 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2001-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The change in psychotic symptoms as measured by Positive and Negative Symptom Scale (PANSS) over 4 week period

SECONDARY OUTCOMES:
Abnormal Involuntary Movement Scale at end of trial period
Adverse Symptom Checklist at end of trial period
Simpson Angus Scale at end of trial period
Hormone Measurements at end of four week period
Cognitive Measurements at end of trial period

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni, MBBS, MPM, FRANZCP, PhD, Principal Investigator — Bayside Health / Monash University
Locations (1):
- Bayside Health - The Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Kulkarni J, de Castella A, Fitzgerald PB, Gurvich CT, Bailey M, Bartholomeusz C, Burger H. Estrogen in severe mental illness: a potential new treatment approach. Arch Gen Psychiatry. 2008 Aug;65(8):955-60. doi: 10.1001/archpsyc.65.8.955. PMID 18678800
- See also: Alfred Psychiatry Research Centre — http://www.med.monash.edu.au/spppm/research/aprc/